CLINICAL TRIAL: NCT04967040
Title: A Comparative Study Between Distally Based Sural Artery Flap and Medial Plantar Artery Flap in Reconstruction of Ankle and Foot Defects
Brief Title: Reconstruction of Ankle and Foot Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Shereef, principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-11
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Foot Injury
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 : medial plantar artery flap (Active Comparator)
  Interventions: Procedure: medial plantar artery flap
- group 2 : distally based sural artery flap (Active Comparator)
  Interventions: Procedure: Distally based sural artery flap

INTERVENTIONS:
Procedure: medial plantar artery flap — Medial plantar artery flap is a fasciocutaneous island flap raised from the non-weightbearing instep of the plantar foot. The dominant vascular pedicle of the flap consists of the medial plantar artery and venae comitantes
  Arms: group 1 : medial plantar artery flap
Procedure: Distally based sural artery flap — Distally based sural artery flap is a fascio-cutaneous island flap taken from the posterior aspect of the middle third of the leg and fed by the lower peroneal septo-cutaneous perforators in reverse fashion. Its vascular basis is the close association between the median superficial sural artery and peroneal artery perforators
  Arms: group 2 : distally based sural artery flap

SUMMARY:
Reconstruction of soft tissue defects around the foot and ankle region is a challenging problem for reconstructive surgeons due to the lack of locally available tissues for transposition, the relatively poor skin circulation, and the special structural characteristics of this area, bones and tendons can easily become exposed due to trauma. so foot injuries are often associated with a loss of soft tissues and exposed bones . The plantar skin is thick, with solid anchorage to the deep structures. Therefore, the reconstructive aim is to restore the stability of the foot skin to adapt to weightbearing and to resist shearing forces. In addition, good sensibility should be considered in the reconstruction. Additional considerations the ankle region has great tension during movement, and good stability is required for shoes wearing. The medial plantar flap has been effectively used in the reconstruction of soft tissue defects localized to the plantar foot, forefoot, posterior heel, and ankle in small to medium sized defects . This flap can be transferred to the defect as a proximally or distally pedicled island flap . The distally based sural artery flap frequently used for reconstruction of soft tissue defects of the lower leg, foot and ankle in medium and large sized defects .Fascio-cutaneous flaps are highly effective and easy to perform.

This study is a comparative study designed for assessment of the clinical applications of distally based sural flap versus medial plantar artery flap regarding the size of the defect , operative technique and their outcomes (success and complications) as a reconstructive option for foot and ankle defects.

ELIGIBILITY:
Inclusion Criteria:

Patients aging 5 to 70 years. Defect at the foot and ankle. Defect size (5- 15) cm2.

Exclusion Criteria:

Severe infection. Unhealthy skin of posterior or lateral aspect of leg . Defect more than 15 cm . Injury to vascular pedicle of the aimed flap .

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Difference in functional outcome between group 1 and group 2 | Difference in functional outcome between group 1 and group 2 is measured at 4 months postoperative
  The functional outcomes are graded as excellent, good, and poor. The criteria for excellent results are the survival of the flap without any flap loss and walking without any aids . Survival of the flap with minimum complications and walking with aids are the criteria for good results. A result is considered poor when an alternative reconstructive procedure is considered

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Li X, Cui J, Maharjan S, Lu L, Gong X. Reconstruction of the Foot and Ankle Using Pedicled or Free Flaps: Perioperative Flap Survival Analysis. PLoS One. 2016 Dec 8;11(12):e0167827. doi: 10.1371/journal.pone.0167827. eCollection 2016. PMID 27930679
- [Background] Hamdi MF, Kalti O, Khelifi A. Experience with the distally based sural flap: a review of 25 cases. J Foot Ankle Surg. 2012 Sep-Oct;51(5):627-31. doi: 10.1053/j.jfas.2012.05.029. Epub 2012 Jul 11. PMID 22789482
- [Background] Uygur F, Duman H, Ulkur E, Noyan N, Celikoz B. Reconstruction of distal forefoot burn defect with retrograde medial plantar flap. Burns. 2008 Mar;34(2):262-7. doi: 10.1016/j.burns.2007.02.010. Epub 2007 Jul 20. PMID 17640813